CLINICAL TRIAL: NCT05936788
Title: Comparative Effects of Active Cycle of Breathing Technique and Diaphragmatic Breathing on Pulmonary Function and Sputum Diary After Coronary Artery Bypass Graft
Brief Title: Comparative Effects of ACBT and Diaphragmatic Breathing on Pulmonary Function and Sputum Diary After CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0310
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Breathing Exercises
Keywords: diaphragmatic exercise; pulmonary function test

STUDY DESIGN:
Intervention Model Description: There will be 2 groups i.e. group A will receive active cycle of breathing technique (ACBT) and group B will receive diaphragmatic breathing technique. Spirometer will be used to evaluate pulmonary functions and breathless, cough and sputum scale (BCSS) will be used to evaluate the improvement in sputum diary of patients. The trial will be completed in two days after patients admitted in the ICUs/CCUs and before and after each session, primary and secondary outcomes will be measured for both groups. A
Who Masked: Participant
Masking Description: There will be 2 groups i.e. group A will receive active cycle of breathing technique (ACBT) and group B will receive diaphragmatic breathing technique. Spirometer will be used to evaluate pulmonary functions and breathless, cough and sputum scale (BCSS) will be used to evaluate the improvement in sputum diary of patients. The trial will be completed in two days after patients admitted in the ICUs/CCUs and before and after each session, primary and secondary outcomes will be measured for both groups. A
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle of breathing technique (Experimental): Group A will receive ACBTs with 1 session a day for total 2 days in a week.
  Interventions: Other: Active cycle of breathing technique
- diaphragmatic breathing (Experimental): Group B will receive diaphragmatic breathing for 1 session a day for total 2 days in a week.
  Interventions: Other: diaphragmatic breathing

INTERVENTIONS:
Other: Active cycle of breathing technique — Group A will receive ACBTs with 1 session a day for total 2 days in a week.
  Arms: Active cycle of breathing technique
Other: diaphragmatic breathing — Group B will receive diaphragmatic breathing for 1 session a day for total 2 days in a week.
  Arms: diaphragmatic breathing

SUMMARY:
To compare the effects of active cycle of breathing technique and diaphragmatic breathing on pulmonary functions and sputum diary after coronary artery bypass graf

DETAILED DESCRIPTION:
It will be a randomized clinical trial. Age of selected subjects will be between 40 to 60 years and data will be collected from intensive care units (ICUs) and cardiac care units (CCUs) of selected hospitals. There will be 2 groups i.e. group A will receive active cycle of breathing technique (ACBT) and group B will receive diaphragmatic breathing technique. Spirometer will be used to evaluate pulmonary functions and breathless, cough and sputum scale (BCSS) will be used to evaluate the improvement in sputum diary of patients. The trial will be completed in two days after patients admitted in the ICUs/CCUs and before and after each session, primary and secondary outcomes will be measured for both groups. After data collection, data will be analyzed using SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

* Post-CABG patients
* Gender: males and females
* Have speaking, hearing and cognitive ability
* On mechanical ventilation for ≤ 24 h after CABG

Exclusion Criteria:

* Prior history of open heart surgery
* Prior severe pulmonary/hepatic or renal disease- Complications after CABG (cardiogenic shock, bleeding requiring transfusion, acute kidney injury, cardiac temponade and severe hypotension)
* Life-threatening arrhythmias (ventricular fibrillation, ventricular tachycardia, atrial fibrillation)
* On mechanical ventilator for more than 24 h after CABG
* Pulmonary complications (atelectasis, acute respiratory distress syndrome (ARDS), diaphragmatic injury)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
6 Min walk test | 4 weeks
  The 6 min walk test is a sub-maximal exercise test used to assess aerobic capacity and endurance.It is also use to monitor your response to treatments for heart lung and other health problems. Provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.

SECONDARY OUTCOMES:
Borg Rating of Perceived scale | 4 weeks
  Is a way of measuring physical activity intensity level.It has a range from 6 to 20 ,scale correlates with a person heart rate or how hard they feel they are working.Ask you to rate the difficulty of your breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Sadiq Saadiq hospital Gujranwala, DHQ hospital Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jasani N, Awad NT, Raut C. Effect of Coronary Artery Bypass Grafting Surgery on Pulmonary Function Tests and Arterial Blood Gases. Indian J Chest Dis Allied Sci. 2016 Jul;58(3):161-164. PMID 30152648
- [Background] Urell C, Westerdahl E, Hedenstrom H, Janson C, Emtner M. Lung Function before and Two Days after Open-Heart Surgery. Crit Care Res Pract. 2012;2012:291628. doi: 10.1155/2012/291628. Epub 2012 Aug 8. PMID 22924127
- [Background] Ono M, Serruys PW, Hara H, Kawashima H, Gao C, Wang R, Takahashi K, O'Leary N, Wykrzykowska JJ, Sharif F, Piek JJ, Garg S, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Noack T, Davierwala PM, Mohr FW, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. 10-Year Follow-Up After Revascularization in Elderly Patients With Complex Coronary Artery Disease. J Am Coll Cardiol. 2021 Jun 8;77(22):2761-2773. doi: 10.1016/j.jacc.2021.04.016. PMID 34082905
- [Background] Moradian ST, Najafloo M, Mahmoudi H, Ghiasi MS. Early mobilization reduces the atelectasis and pleural effusion in patients undergoing coronary artery bypass graft surgery: A randomized clinical trial. J Vasc Nurs. 2017 Sep;35(3):141-145. doi: 10.1016/j.jvn.2017.02.001. PMID 28838589
- [Background] Montrief T, Koyfman A, Long B. Coronary artery bypass graft surgery complications: A review for emergency clinicians. Am J Emerg Med. 2018 Dec;36(12):2289-2297. doi: 10.1016/j.ajem.2018.09.014. Epub 2018 Sep 8. PMID 30217621
- [Background] Rademacher J, Welte T. Bronchiectasis--diagnosis and treatment. Dtsch Arztebl Int. 2011 Dec;108(48):809-15. doi: 10.3238/arztebl.2011.0809. Epub 2011 Dec 2. PMID 22211147